CLINICAL TRIAL: NCT01508078
Title: Characterization of Adult Subjects for Asthmatic Research Studies
Acronym: CASA
Status: Suspended | Type: Observational
Why Stopped: The restrictions on research imposed for the COVID-19 pandemic prevented us from continuing recruitment and visits. At this stage our funding is not sufficient to continue enrollment so we will put the study in a hold pattern.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 10-01627
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of induced sputum and blood for DNA and RNA extraction, plasma, and serum will be banked in the UCSF Airway Tissue Bank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthmatics: Otherwise healthy asthmatic subjects
- Healthy controls: Healthy individuals without evidence of pulmonary disease.

SUMMARY:
This study is designed to characterize subjects in terms of the nature and severity of their asthma and in terms of conditions that may alter the clinical expression of asthma. Some features will be obtained in all subjects. These include a medical history and baseline lung function tests. This characterization forms the basis for our database that facilitates research protocols.

DETAILED DESCRIPTION:
The purpose of this study is to generate a cohort of well-characterized asthmatic subjects as a resource for recruitment of asthmatic subjects and healthy controls in clinical studies and clinical trials in the UCSF Airway Clinical Research Center. The UCSF Airway Clinical Research Center (ACRC) conducts multiple clinical research studies in asthma funded by the NIH, foundations, and industry. We have a broad range of research interests, but we have specific interests in mechanism-oriented clinical studies and specific expertise in biospecimen collection, biobanking, and biospecimen analysis. Our model is to have multiple studies recruiting simultaneously, and this means that we need well-organized recruitment and database systems.

Additionally, we aim to characterize asthmatic subjects in multiple domains, including disease severity, airway inflammation subtypes, and mucus subtypes. Asthma is a heterogeneous disease in its clinical presentation and in its underlying cellular and molecular phenotypes. To explore cellular and molecular phenotypes of asthma, we will analyze induced sputum for cell types and gene expression, with a focus on Th2 inflammation pathways and innate and adaptive immune cells that drive Th2 inflammation. Detailed cellular analysis of sputum is possible but requires that multiple sputum samples be collected for processing in multiple different ways, including by cytocentrifugation, FACS analysis, and by formalin fixation and paraffin embedding of sputum cell pellets. We are also studying mucus phenotypes of asthma using methods of rheology, which needs to be done on fresh sputum.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older

Exclusion Criteria:

* History of lung disease other than asthma
* An upper respiratory tract infection or an exacerbation of their asthma within the preceding 4-6 weeks.
* Persons who have smoked > 5 cigarettes per month and have a total pack-year smoking history > 10 packs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthmatics and healthy control
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Airway inflammation | Cross-sectional
  We will measure various indicators of airway inflammation and compare them with various phenotypic characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- See also: Airway Clinical Research Center website — http://acrc.ucsf.edu